CLINICAL TRIAL: NCT06729229
Title: The YOU-Fish Study: Exploring the Effects of Fish Consumption and Omega 3 Supplementation on the Vascular Health of Young Adults
Brief Title: The YOU-Fish Study: Fish and Omega 3 Supplementation in Young Adults
Acronym: YOU-Fish
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: REC/24/0005
Record Dates: First submitted 2024-11-15; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Prevention
Keywords: Polyunsaturated fatty acids; Omega 3 index; fish, fish consumption; cardiovascular disease.
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dietary Supplements; Vitamins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fish and Placebo (Experimental): Participants will receive 2 portions of fish (280g)
  Interventions: Dietary Supplement: Placebo
- No fish SUPPLEMENT (Experimental): Daily 1g omega-3 supplement
  Interventions: Dietary Supplement: Dietary Supplement/Vitamins
- No fish PLACEBO (Experimental): Placebo
  Interventions: Dietary Supplement: Placebo
- 2 fish portion (Experimental): Omega 3 supplement
  Interventions: Dietary Supplement: Dietary Supplement/Vitamins

INTERVENTIONS:
Dietary Supplement: Placebo — Experimental - 2 portions of fish (280g) per week and placebo supplement (corn oil)
  Arms: Fish and Placebo
Dietary Supplement: Dietary Supplement/Vitamins — Experimental - Control lunch (no fish) and omega 3 supplement
  Arms: 2 fish portion
Dietary Supplement: Placebo — Placebo comparator - Control lunch (no fish) and placebo supplement
  Arms: No fish PLACEBO
Dietary Supplement: Dietary Supplement/Vitamins — Experimental - 2 portions of fish (280g) per week and omega 3 supplement
  Arms: No fish SUPPLEMENT

SUMMARY:
Cardiovascular disease (CVD) is one of the major causes of mortality, however, it is estimated that approximately 75% of all cases are preventable. Previous evidence has shown higher blood concentrations of n-3 polyunsaturated fatty acids (PUFAs) are associated with a lower risk of cardiovascular disease owing to their ability to lower inflammation. The omega-3 index (O3I) is a commonly used marker of n-3 PUFA status, which refers to the percentage of n-3 long chain PUFAs (with respect to total fatty acids) in red blood cell membranes, with an O3I of >8% associated with the lowest risk of CVD. Concerningly it's estimated that most of the population have an O3I ranging from 4-5%. Fish is a rich source of polyunsaturated fatty acids (PUFA) and has been shown to be one of the main predictors of a higher O3I. Current guidelines recommend the consumption of 2 portions of fish per week; however, current UK and Irish intakes are well below the current recommendations, particularly amongst young people. Additionally, professional bodies have noted that a daily omega-3 supplement, providing approximately 500mg EPA + DHA per day, is beneficial in increasing omeag-3 intakes amongst those who may exclude dietary sources such as fish. The regular consumption of fish or omega 3 supplement use could help to increase the O3I, however, it remains unknown as to whether the guidance surrounding these methods are effective in reaching the recommended target of 8%. Early interventions such as increasing the O3I (throughfish and/or supplements) into a lower risk category may be an effective intervention in the prevention of CVD. This human intervention study will investigate the effects of omega 3 supplements and fish on the O3I and vascular health of young adults. It is hypothesised that increasing fish consumption or taking omega 3 supplements will increase the O3I and improve the vascular health of young adults.

DETAILED DESCRIPTION:
Apparently healthy males and females aged between 18-30 years old and who are low consumers of fish and not regularly consuming fish oil, or protein supplements will be recruited. A blood spot will be taken as part of the screening process to ensure the participants have a low baseline O3I (less than 6%) and to confirm they are low fish consumers and are not taking any supplements containing n-3 PUFA. A 2x2 factorial design will explore the effects of consuming fish and omega-3 supplements on the O3I and health of young adults. Participants will be randomly allocated, by an independent researcher, to one of 4 intervention groups: (I) a fish meal and omega-3 supplement group, (ii) a fish meal and placebo supplement group, (iii) a control meal (no fish) and omega-3 supplement, or (iv) a control meal (no fish) group and placebo supplement. Participants in the dietary fish group will be asked to attend the HISU twice per week where they will receive two lunch dishes per week containing a total of 280g fish per week (based on SACN dietary advice, SACN, 2004) for 8 weeks (140g oily fish and 140g lean fish) whilst the participants in the control group will receive a control meal. Examples of fish lunches may include salmon with a side of salad or a fish pie. Participants allocated to receive a control meal will be asked to attend the HISU at Ulster University where they will be provided with a fish free lunch such as cottage pie or chicken with a side of salad. The PUFA composition of the fish will be determined.

Participants in the omega-3 supplement or the placebo control group will be asked to consume a daily 1g omega-3 supplement (400mg EPA + 200mg DHA) or a daily 1g control capsule for 8 weeks, respectively. The control capsules will contain corn oil to deliver a fatty acid composition similar to that of the UK diet. Participants will be blinded as to whether they have been allocated supplements or placebo control which will be flavoured with peppermint and asked to take the supplement during a high fat meal (e.g. dinner) to enhance bioavailability and reduce intervariability amongst participants.

Participants will be asked to attend a baseline and post intervention appointment at the HISU at Ulster University. Body height (stadiometer), weight and composition (TANITA scales) will be determined. A fasting blood sample and faecal sample will be obtained and stored until batch analysis. The study will investigate the impact of fish and omega-3 supplements on the omega-3 index (OmegaQuant), full lipid profile (Daytona clinical analyser), full blood profile and immune markers related to cardiovascular disease such as c-reactive protein (CRP) and tumour necrosis factor alpha (TNF-α), interferon gamma (IFN-γ) and interleukins (IL-1β, IL-2, IL-4, IL-6, IL-10) using validated immunoassays, and gut microbiota.

Participants will be invited to partake in a short focus group (lasting approximately 1 hour) and complete a short questionnaire at baseline and 8 weeks post intervention to ascertain consumer attitudes (knowledge, awareness, behaviours, and barriers) towardsfish consumption and supplement use and how these have changed as a result of completing the intervention study.

All statistical analyses will be completed per protocol and using intention-to-treat (ITT) analyses. The primary analysis will compare (1) all those randomised to the fish intervention versus all those not allocated to the fish intervention and (2) all those randomised to the omega-3 supplement versus all those not allocated to the omega-3 supplement. Analysis of covariance controlling for age, BMI, and baseline O3I will be used to determine the effect of the interventions.

In a fixed effects ANOVA (comparison of means), sample sizes of 5 in each of the 4 groups (20 in total) achieves 91% power to detect a difference of 2.0% in O3I change using the Tukey-Kramer (Pairwise) multiple comparison test at a 0.05 significance level. A higher number of participants tend to drop out post randomisation before starting the intervention and this tends to exceed the expected 10% drop out rates and result in an attrition rate closer to 20%. Given the lower sample size needed and the risk of potential dropouts, in order to ensure the required 5 participants complete each of the 4 treatment groups, 10 participants will be recruited per group leading to a total sample size of 40.

ELIGIBILITY:
Inclusion Criteria:

* Omega 3 index <6% Healthy males or females.
* Aged 18-30 years old.
* Low consumers of fish (<2 portions/month).
* Willing to 2 portions (280 grams) of fish per week.
* Not consuming fish oil supplements.
* Not consuming protein supplements.
* Within a BMI of 18-30kg/m2
* Not allergic to seafood

Exclusion Criteria:

* Omega 3 index >6%
* Regularly consume fish.
* Are allergic to seafood.
* Are taking fish oil supplements (for example fish oil, cod oil, krill oil, GLA or evening primrose) or are taking protein supplements (for example whey protein).
* Are pregnant/lactating.
* Have existing health conditions such as Diabetes Mellitus and known hypertension.
* Dietary restrictions resulting in the exclusion of fish such as vegan.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males and females will be recruited
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Omega 3 index measured as percentage | Change at 8 weeks from baseline
  Assessed via Gas-Chromatography mass spectrometry

SECONDARY OUTCOMES:
Polyunsaturated fatty acid status | Time frame: change at 8 weeks from baseline
  mg/ml

OTHER OUTCOMES:
Inflammatory status | Change at 8 weeks from baseline
  Cytokine concentration pg/ml
Lipid Profile | Change at 8 weeks from baseline
  Serum Lipid profile mmol/l
Microbiota | Change at 8 wees from baseline
  Faecal microbiota profile % relative abundance

CONTACTS AND LOCATIONS:
Overall Officials: Emeir McSorley, PhD, Principal Investigator — Ulster University, Cromore Road, Coleraine, Co. Londonderry, BT521SA.
Locations (1):
- NICHE, School of Biomedical Sciences, Biomedical Sciences Research, Coleraine Campus, University of Ulster, Coleraine, Co Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McMullan JE, Kumar RA, Yeates AJ, Allsopp PJ, Mulhern MS, van Wijngaarden E, Strain JJ, McSorley EM. Influence of Fish Consumption and omega-3 Supplementation on the omega-3 Index of Young Adults: A 2 x 2 Factorial Randomized Controlled Trial (YouFish Study). J Nutr. 2025 Dec;155(12):4345-4355. doi: 10.1016/j.tjnut.2025.10.010. Epub 2025 Oct 11. PMID 41082976